CLINICAL TRIAL: NCT06662578
Title: Exploring Neurocognitive Stimulation in Dementia Through Equine-Assisted Therapy: A RCT Pilot Study
Brief Title: Using Equine Therapy in Dementia Cognitive Stimulation
Acronym: ETMW_DEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Responsible Party: Principal Investigator, Madeline Alford, Master's student, Cooperativa de Ensino Superior, Politécnico e Universitário
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 05/CE-UICS/2024
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Dementia
Keywords: Dementia; Equine therapy; Neurocognitive stimulation; Memory workshop; Quality of life; Alzheimer's; Depression
MeSH Terms: conditions — Dementia; Depression | interventions — Animal Assisted Therapy; Equine-Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention)
- Traditional memory workshop (Active Comparator): Neurocognitive stimulation as usual
  Interventions: Other: Traditional memory workshop
- Equine assisted therapy memory workshop (Experimental): Neurocognitive stimulation mediated with a horse based on a defined protocol.
  Interventions: Other: Equine assisted therapy memory workshops

INTERVENTIONS:
Other: Traditional memory workshop — The participants received 8 weekly sessions of 60 minutes of neurocognitive stimulation, based on French memory workshops.
  Other Names: neurocognitive stimulation; cognitive stimulation; memory workshops
  Arms: Traditional memory workshop
Other: Equine assisted therapy memory workshops — The participants received 8 weekly sessions of 60 minutes, based on traditional memory workshops (French type of neurocognitive stimulation) with the mediation of a horse (example : working on associative memory by selecting which object is used for the horse between 2 presented objects).
  Other Names: Animal assisted therapy; Equine therapy; neurocognitive stimulation; Equine mediation
  Arms: Equine assisted therapy memory workshop

SUMMARY:
The goal of this clinical trial is to learn if integrating equine therapy in memory workshops in mild to moderate Dementias can improve cognitive function, quality of life and mood. The main question[s] it aims to answer is:

Does the mediation of a horse in memory workshops increase its effects ?

Researchers will compare traditional memory workshops, memory workshops using equine therapy and a control group to see if the equine therapy mediation will increase cognitive functions, mood and quality of life in individuals with mild to moderate Dementias.

Participants will participate in 8 weekly sessions of equine therapy memory workshops / traditional memory workshops / a control group will not have any interventions during that period. All subjects will be evaluated pre and post intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Have been medically diagnosed with Major Neurocognitive Disorders
* Scores between 0.5 and 2 on the Cognitive Dementia Rating scale (CDR) (Berg, 1982)
* Adults of all genders, aged 65 and over; and
* Willingness to participate in a memory workshop; e) willingness to interact with a horse.

Exclusion Criteria:

* Expressed fear, aversion, or has had a negative experience with horses
* Allergy or other medical condition which did not allow contact with horses.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function as Assessed by the Montreal Cognitive Assessment (MoCA) | Baseline and ten weeks after
  Pre and post-intervention period, the Montreal Cognitive Assessment was used to assess cognitive function.

SECONDARY OUTCOMES:
Change in Depression Symptoms as Assessed by the Geriatric Depression Scale (GDS-15) | Baseline and ten weeks after
  Assessment of depression levels pre and post-intervention using the Geriatric Depression Scale - 15 items
Change in Quality of Life as Assessed by the Quality of Life in Alzheimer's Disease (QoL-AD NH) | Baseline and ten weeks after
  Assessment of the quality of life pre and post intervention using the Quality of life in Alzheimer's Disease - Nursing homes .

CONTACTS AND LOCATIONS:
Locations (1):
- CAJOU, Le Boulou, France

IPD SHARING:
Plan to Share IPD: No